CLINICAL TRIAL: NCT05696327
Title: Effects of Eccentric Tyler Twist Extensor Strengthening Exercises in Lateral Epicondylitis
Brief Title: Eccentric Tyler Twist Wrist Extensor Strengthening in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Riphah/RCRS/01222 Rimsha Jalil
Record Dates: First submitted 2023-01-04; First posted 2023-01-25 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis, Tyler Twist Exercises, Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): tyler twist wrist extensor strengthening exercises Treatment protocol will be followed for thrice a week for 4 weeks. The session will be of approximately 20 minutes. The initial Conventional therapy program will be the same as discussed in the control group except strengthening exercise which is excluded in experimental group because of Tyler twist exercise which is being used as a strengthening protocol.
  Interventions: Other: Tyler Twist Exercises
- Control Group (Active Comparator): Conventional physiotherapy (Ultrasound + Cross Friction Massage for 10 minutes + Wrist extensor stretching and Isotonic wrist extensor strengthening.) The treatment will continue for 4 weeks and 3 sessions/ week i.e. thrice a week. The session will be of approximately 20 minutes.
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: Tyler Twist Exercises — Tyler twist exercises are the group of exercises which are used to strengthen wrist ex tensors.The protocol consists of several steps using colored twist-able bands and patients are guided to actively perform the steps for their grip strength development.
  Arms: Experimental Group
Other: conventional physical therapy — Conventional physiotherapy (Ultrasound + Cross Friction Massage for 10 minutes + Wrist extensor stretching and Isotonic wrist extensor strengthening.)
  Other Names: control group
  Arms: Control Group

SUMMARY:
The purpose of the study is to compare the effects of Tyler twist wrist extensor strengthening exercises in patients with lateral epicondylitis. A randomized control trial was conducted at Cina medical center Rawalpindi and Midland Doctors Medical institute. The sample size was 52 calculated through open-epi tool. The participants were divided into two groups: the treatment group and the control group. The study duration was 1 year. Sampling technique applied was non-probability purposive sampling. Only 20 to 40 years participants with diagnosed condition were included in the study. Tools used in this study are Jamar dynamometer for grip strength and PRTEE Questionnaire for pain and disability. Data was collected at baseline, mid and immediately after the application of interventions. Data analyzed through SPSS version 25

DETAILED DESCRIPTION:
Lateral epicondylitis is the most common cause of pain in elbow, due to repetitive wrist extension or gripping activities. This condition is also described as a chronic symptomatic degeneration of the extensor tendon of forearm commonly extensor carpi radialis brevis at the attachment area of humeral epicondyle. (1) Tennis elbow is common in individuals who undergo repetitive wrist extension, radial deviation, and forearm supination. The histological findings of lateral epicondylitis consist of granulation tissue, micro-rupture, fibroblasts abundance, UN structured collagen, vascular hyperplasia, and lack of inflammatory cells within the tissue (lymphocytes, macrophages, neutrophils). (2) Lateral epicondylitis can occur in any age group but is more common between 30-50 years of age. (3) Many previous reports conducted in different countries described that there is 2-14% prevalence of lateral epicondylitis in working population and only 5% of people suffering from tennis elbow relate this injury to the tennis. (4) Evidence from a systematic review published in 2019 described the prevalence rate of 1-3% in the general population and 7% in the handy workers group with equal gender distribution. (5) There are many treatment options for lateral epicondylitis. Initially it is treated by conservative treatment (1) Recently in 2021, R Manandhar et al conducted an RCT reported positive results using combination of Movement with mobilization and Eccentric exercises regarding pain and functional disability.(8) BL Woodley et al in 2018 published his systematic review which concluded that limited level of evidence exists on the effectiveness of eccentric strengthening exercises to standard physiotherapy protocols. Twenty relevant studies were sourced, 11 of which met the inclusion criteria. These included studies of tendinopathy of the common wrist extensor tendon of the lateral elbow (LET. (9) If pain do not resolve with conservative treatment then further treatment options will be extracorporeal shock wave therapy, cortisone injections and surgery.(6) In an RCT of Ju-hyun Lee et all in 2018 ,the effects of eccentric control exercise for tennis elbow showed useful effects for pain and functional activity was improved with a p value of 0.05.(7) Timothy Tyler et al recently conducted a cross sectional study in 2021 to compare standard physiotherapy treatment to Tyler twist exercises which are a new treatment protocol for wrist extensor strengthening using 2-3 colored twistable rubber bands This study suggested that Tyler twist exercise could be effective strength training protocol and once learnt can be performed by the patient at home without any supervision.(9)

To treat lateral epicondylitis platelet rich plasma has gained popularity. To enhance wound healing, bone healing and tendon healing, platelets release high concentration of platelet-derived growth factors. It is difficult to draw clear conclusions on PRP for lateral epicondylitis because some available studies have reported conflicting results. Manipulative techniques fall into two basic varieties in the treatment of lateral epicondylitis; those that will produce a thrust and those that seek full extension. To effect the contractile element the manipulations performed in extension with pronation have the greatest chance. Forced extension of elbow with the wrist and fingers fixed and the forearm promoted is the most common procedure known as mill's manipulation. Manipulations are painful procedures and require 2 weeks of rest after application.(11) With a high success rate, injections are one of the most popular methods utilized .Physical therapy is initiated when the condition becomes chronic or not responding to initial treatment. Ultrasound, phonophoresis, electrical stimulation,, manipulation, soft tissue mobilization , neural tension, friction massage , augmented soft tissue mobilization and stretching and strengthening techniques are the common rehabilitation modalities utilized for the treatment. (12) Proper evidence behind Tyler twist wrist extensor exercises in the management of lateral epicondylitis is sparse and there are less number of studies with limited methodological designs. There are no previous randomized control trials conducted to see the effects of Tyler twist exercises in contrast to standard physiotherapy treatment using combined tools for pain , grip strength and functional activity According to the literature review, there had been lack of reporting of compliance and adherence to the exercise programs, with only four studies documenting exercise adherence, So, the additional benefit of this protocol is that it can be performed as part of a home program and does not involve continued medical supervision when learned properly. So, this study will focus on effects of Tyler twist exercise to standard physiotherapy protocol.

ELIGIBILITY:
Inclusion Criteria:

* both genders (male and female)
* Age between 20yrs-40yrs
* Tenderness on palpation over the lateral epicondyle of humerus.
* Pain with gripping.
* Pain with resisted wrist extension.
* clinically diagnosed patients of lateral epicondylitis
* did not take any kind of physiotherapy treatment.

Exclusion Criteria:

cervical spine disorder.

* Peripheral neuropathy.
* Previous Fracture/ trauma or surgery to the elbow region.
* Steroid injections in last 6 months.
* Tumor or wound.
* Any other systemic/autoimmune disorders or congenital Participants who received any therapy for lumbar region past 3 days

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Hand held dynamo-meter(Grip strength) | upto 24 weeks
  To measure grip strength, Hand held dyanamo-meter is used as a tool to record readings in Kg.The device is hand held and displays grip force with a maximum range of 90kg.Maximum 3 readings are recorded and then a mean is calculated which is an actual value to be noted.Male to female ratio varies for the grip strengths and ranges from 35kg max in females and 60kg in male population.Strength also varies in old population as well.

SECONDARY OUTCOMES:
Patient rated tennis elbow evaluation questionnaire(PRTEE) | upto 24 weeks
  Pain and disability are the two variables which are measured using PRTEE(Patient rated tennis elbow evaluation questionnaire). The questionnaire consists of 3 portions :(Pain , Functional disability usual activities and functional disability specific activities ,Total score ). To measure forearm pain and disability , this 15 item assessment tool is used to record the readings(Baseline , mid and post interventional assessments) .

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No